CLINICAL TRIAL: NCT03796325
Title: Effect of Laparoscopic Sleeve Gastrectomy in Obese Patients With Depressive State
Brief Title: Depressive State After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of the Department of General Surgery, Assuta Medical Center
Other Study IDs: AMC 002-2018
Record Dates: First submitted 2018-12-29; First posted 2019-01-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Morbid; Depression
MeSH Terms: conditions — Obesity, Morbid; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Depression: patients characterize with morbid obesity or obesity type 2 with co-morbidities and depression
- No-depression: patients characterize with morbid obesity or obesity type 2 with co-morbidities without depression

SUMMARY:
Obesity is an epidemic disease that continues to increase causing morbidity and mortality to those who suffer. Obese patients suffer, frequently, from a depressive state, anger, and emotional disturbances. It cannot be recognized and depression causes obesity affecting eating habits or obesity causes depression based on physical, social and occupational limitations. Many times we see that obese patients are discriminated in every sense of daily life increasing their depressive state. The best treatment for obesity is bariatric surgery that causes a sufficient weight loss to correct sleep apnea, diabetes, hypertension, and many other co-morbidity. The study is based on elucidating the effect of sleeve gastrectomy in obese patients suffering from depression

DETAILED DESCRIPTION:
The patients were classified as suffering from a depressive state before the bariatric surgery and followed until 3 years after surgery, the data was collected by personal interview or telephone survey.

ELIGIBILITY:
Inclusion Criteria: 18 years and older No any type of complication after surgery No difficult to drink, eat or take medicaments

Exclusion Criteria:

Any surgical complication Previous gastrointestinal surgery schizofrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older with BMI at less 40 or 35-40 with co-morbidities
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Weight loss 3 years after laparoscopic sleeve gastrectomy | 36 month
  Measure of weight calculating Delta body mass index between preoperative measurement and three years after surgery

SECONDARY OUTCOMES:
Depression state changes after Sleeve gastrectomy | 36 month
  Telephonic Questionnaire about feeling satisfaction (Very satisfied, satisfied, indifferent ,unsatisfied), eating mode (Volume-eater, sweet-eater, snack eater, binge eater, healthy-eater), occupations (Unemployed, employed, type of employment).

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta MC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Griauzde DH, Ibrahim AM, Fisher N, Stricklen A, Ross R, Ghaferi AA. Understanding the psychosocial impact of weight loss following bariatric surgery: a qualitative study. BMC Obes. 2018 Dec 3;5:38. doi: 10.1186/s40608-018-0215-3. eCollection 2018. PMID 30524743